CLINICAL TRIAL: NCT02059668
Title: Observational Study on Biomarkers in Head and Neck Cancer
Brief Title: Observational Study on Biomarkers in Head and Neck Cancer (HNprädBio)
Acronym: HNprädBio
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Prof. Dr. Mechthild Krause, Technische Universität Dresden
Other Study IDs: STR- HNprädBio-2013
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer
Keywords: locally advanced head and neck cancer; biomarkers; definitive treatment; adjuvant treatment; radiochemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — if possible fresh-frozen tumor tissues, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomarker analyses head & neck cancer tissue, blood specimen: Validation of prognostic biomarkers for local tumor control in definitive and adjuvant treatment of head and neck cancer.
  Interventions: Biological: Biomarker analyses head & neck cancer tissue, blood specimen

INTERVENTIONS:
Biological: Biomarker analyses head & neck cancer tissue, blood specimen — For biomarker analyses, tumor tissues from previous biopsies and surgery and blood specimens taken during treatment at the treating institution will be used.

SUMMARY:
The aim of this clinical research project is to validate the prognostic impact of potential biomarkers on loco-regional control of locally advanced head and neck cancer after definitive or adjuvant radiochemotherapy. The treatment is equal to the standard of care.

Potential biomarkers from a previous retrospective study will be validated in this prospective study.

DETAILED DESCRIPTION:
Objectives:

Primary: Evaluation of local-regional recurrence- free survival after two years of patients with locally advanced head and neck cancer who received definitive or adjuvant radiochemotherapy.

Secondary: Evaluation of disease-free -survival, metastases-free and overall survival after two years, of patients with locally advanced head and neck cancer.

Outline: This is a multicenter observational study. The treatment is based on the center specific standard of care. The total dose will be between 69 and 73 Gy (definitive treatment) and 63 and 66 Gy (adjuvant treatment), the chemotherapy will be cisplatin- based.

The aim of the analysis is to validate the prognostic impact of potential biomarkers on loco-regional control. This will lead to the definition of risk groups and stratification of patients and will help to individualize radiotherapy prescription in future trials.

ELIGIBILITY:
Inclusion Criteria:

Primary radiochemotherapy:

* Patients with locally advanced squamous cell carcinoma of the oral cavity, oropharynx or hypopharynx
* Stage III or IV without distant metastases
* Patient is able to participate in regular tumor follow-up care
* planned irradiation dose 69-72 Gy
* planned overall treatment time 38-54 days
* written informed consent of the patient
* general condition according to WHO 0-2
* planned simultaneous chemotherapy with cisplatin (cumulative planned total dose minimum 180 mg/m2 body surface, divided in several separately doses)

Adjuvant radiochemotherapy:

* Patients with locally advanced squamous cell carcinoma of the oral cavity, oropharynx or hypopharynx
* surgery, existence of one or more of the following risk factors for local recurrence:
* extracapsular growth of a minimum of one lymph node metastasis
* R1 resection
* pT4 tumor and more than 3 affected lymph nodes
* Patient is able to participate in regular tumor follow-up care
* planned irradiation dose 63-66 Gy
* planned overall treatment time 44-48 days
* planned simultaneous chemotherapy with cisplatin (cumulative planned total dose minimum 200 mg/m2 body surface, divided in several separately doses)
* written informed consent of the patient
* general condition according to WHO 0-2
* time since last surgery <56 days (8 weeks)

Exclusion Criteria:

Primary radiochemotherapy:

* distant metastasis
* contraindication against a cisplatin-based chemotherapy
* planned total irradiation dose <69 Gy and >72 Gy
* planned overall treatment time >54 days or <38 days
* Patient is incapable of giving consent
* previous radiotherapy in the head and neck area, if there is a risk for overlapping of the irradiation areas
* other tumor diseases, which currently need a treatment or probably within the next two years or which influence the prognosis of the patient
* tumor-independent diseases or conditions which reduce the survival probability of the patient to <2 years or which affect the follow-up over 2 years
* no written informed consent
* induction chemotherapy
* pregnancy or lactation

Adjuvant radiochemotherapy:

* distant metastasis
* contraindication against a cisplatin-based chemotherapy
* planned total irradiation dose < 63 Gy or > 66 Gy
* planned overall treatment time > 48 days or < 44 day
* Patient is incapable of giving consent
* previous radiotherapy in the head and neck area, if there is a risk for overlapping of the irradiation areas
* other tumor diseases, which currently need a treatment or probably within the next two years or which influence the prognosis of the patient
* tumor-independent diseases or conditions which reduce the survival probability of the patient to <2 years or which affect the follow-up over 2 years
* no written informed consent
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis locally advanced squamous cell carcinoma of the head and neck area
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2014-03; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
local recurrence free survival | after 2 years

SECONDARY OUTCOMES:
disease-free survival | after 2 years
metastases-free survival | after 2 years
overall survival | after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Principal Investigator — Dresden University of Technology, Universital Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology
Locations (10):
- Germany (10):
  - Prof. Anca-Ligia Grosu, Freiburg im Breisgau, Baden-Wurttemberg
  - Prof. Jürgen Debus, Heidelberg, Baden-Wurttemberg
  - Prof. Daniel Zips, Tübingen, Baden-Wurttemberg
  - Prof. Claus Belka, München, Bavaria
  - Prof. Stephanie Combs, München, Bavaria
  - Prof. Claus Rödel, Frankfurt am Main, Hesse
  - Prof. Martin Stuschke, Essen, North Rhine-Westphalia
  - Prof. Mechthild Krause, Dresden, Saxony
  - Prof. Volker Budach, Berlin
  - Praxis für Strahlentherapie im Krankenhaus Dresden - Friedrichstadt, Dresden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niu M, Combs SE, Linge A, Krause M, Baumann M, Lohaus F, Ebert N, Tinhofer I, Budach V, von der Grun J, Rodel F, Grosu AL, Multhoff G. Comparison of the composition of lymphocyte subpopulations in non-relapse and relapse patients with squamous cell carcinoma of the head and neck before, during radiochemotherapy and in the follow-up period: a multicenter prospective study of the German Cancer Consortium Radiation Oncology Group (DKTK-ROG). Radiat Oncol. 2021 Jul 31;16(1):141. doi: 10.1186/s13014-021-01868-5. PMID 34332614